CLINICAL TRIAL: NCT01768091
Title: Peroral Endoscopic Myotomy Versus Pneumatic Dilation for Esophageal Achalasia: a Prospective Randomized Controlled Trial
Brief Title: POEM vs. Pneumatic Dilation for Esophageal Achalasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-201211-K2; 201120 (Other Grant/Funding Number: New business and New Technology Project of Nanfang Hospital)
Record Dates: First submitted 2013-01-05; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Esophageal Achalasia
Keywords: Esophageal achalasia; Peroral endoscopic myotomy; POEM; Pneumatic dilation
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POEM (Experimental): POEM for patients with esophageal achalasia
  Interventions: Procedure: POEM
- Pneumatic dilation (Active Comparator): Pneumatic dilation for patients with esophageal achalasia
  Interventions: Procedure: Pneumatic dilation

INTERVENTIONS:
Procedure: POEM — 1. Entry to submucosal space. After submucosal injection, a 2-cm longitudinal mucosal incision is made at approximately 13 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnelling. A long submucosal tunnel is created to 3 cm distal to the GEJ.
  3. Endoscopic myotomy is begun at 3 cm distal to the mucosal entry point, and is carried out in a proximal to distal direction to a total length of 10 cm.
  4. Long endoscopic myotomy of inner circular muscle bundles is done, leaving the outer longitudinal muscle layer intact. The expected end point of myotomy is 2 cm distal to the GEJ.
  5. Closure of mucosal entry: the mucosal incision is closed using hemostatic clips.
  (Inoue H et al. POEM for esophageal achalasia… Endoscopy 2010; 42: 265-271)
  Other Names: Peroral endoscopic myotomy
  Arms: POEM
Procedure: Pneumatic dilation — A Rigiflex balloon (30 mm) was positioned at the esophagogastric junction and dilated at a pressure of 5 PSI for 1 minute, followed by 8 PSI for 1 minute.
  (N Engl J Med 2011;364:1807-16.)
  Arms: Pneumatic dilation

SUMMARY:
The purpose of this study is to determine the efficacy and safety of peroral endoscopic myotomy (POEM) compared with pneumatic dilation in the treatment of esophageal achalasia.

DETAILED DESCRIPTION:
Esophageal achalasia is an esophageal motor disorder, which is characterized by the absence of esophageal peristalsis combined with a defective relaxation of the lower esophageal sphincter (LES). The major symptoms of esophageal achalasia are dysphagia, chest pain, and regurgitation of undigested food.

Currently, treatment options mainly focus on relief of the symptoms by reducing the LES pressure. Pneumatic dilation is the main endoscopic therapies for esophageal achalasia. However, the patients need repeat treatment to maintain therapeutic success and there is a risk of perforation (1%-3%). For surgery approaches, the laparoscopic Heller's myotomy (LHM) combined with Dor's antireflux procedure has gained considerable interest. The LHM can sustain therapeutic effects for long-term in approximately 80% of patients.

Recently, Inoue et al. succeeded in treating achalasia endoscopically with a method called peroral endoscopic myotomy (POEM) and achieved promising results in short-term. Technically, POEM derived from natural orifice transluminal endoscopic surgery (NOTES) and endoscopic submucosal dissection (ESD), in which a submucosal tunnel is created after submucosal injection, and then an endoscopic myotomy was made at the gastroesophageal junction.

However, the long-term efficacy and safety of POEM were not determined, and there was no prospective study that compared the POEM with other conventional treatment. Therefore, we aim to determine the efficacy and safety of POEM, compared with the pneumatic dilation, in the treatment of esophageal achalasia.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age
* Patient with esophageal achalasia
* Eckardt score > 3
* Signed informed consent

Exclusion Criteria:

* Severe cardio-pulmonary disease or other serious disease leading to unacceptable surgical risk
* Pseudo-achalasia, Mega-oesophagus (greater than 7 cm), or Oesophageal diverticula in the distal oesophagus
* Previous endoscopic Botox injection
* Previous oesophageal or gastric surgery
* Pregnancy or lactation women, or ready to pregnant women
* Not capable of filling out questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success | From date of randomization until the follow-up ended, assessed up to 2 years
  Therapeutic success is defined as a symptom control to an Eckardt score of 3 or less.
  The Eckardt score is the sum of the symptom scores for dysphagia, regurgitation, and chest pain (with a score of 0 indicating the absence of symptoms, 1 indicating occasional symptoms, 2 indicating daily symptoms, and 3 indicating symptoms at each meal) and weight loss (with 0 indicating no weight loss, 1 indicating a loss of <5 kg, 2 indicating a loss of 5 to 10 kg, and 3 indicating a loss of >10 kg) (Eckardt, V. Gastroenterology, 1992. 103(6): p. 1732-8.)

SECONDARY OUTCOMES:
Procedure related complication | From date of randomization until the follow-up ended, assessed up to 2 years
  Perforation, Delayed bleeding, Pneumothorax, Subcutaneous emphysema, Anastomotic leak etc.
Time of treatment failure | From date of randomization until the follow-up ended, assessed up to 2 years
  Time of treatment failure is defined as when the Eckardt score of patients are more than 3
Pressure at the lower esophageal sphincter | From date of randomization until the follow-up ended, assessed up to 2 years
  The basal LES pressure and the swallow-induced LES relaxation will be monitored and measured at the end of expiration. After introduction and equilibration, basal pressure is monitored during at least 5 minutes. Swallow-induced relaxation of the sphincter is assessed by 5 ml wet swallows, at least 30 s apart.
Quality of life | From date of randomization until the follow-up ended, assessed up to 2 years
  Patients will complete the quality-of-life questionnaires (the Medical Outcomes Study 36-Item Short-Form Health Survey, SF-36) for assessing quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gong, M.D., Principal Investigator — Department of Gastroenterology, Nanfang Hospital of Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Boeckxstaens GE, Annese V, des Varannes SB, Chaussade S, Costantini M, Cuttitta A, Elizalde JI, Fumagalli U, Gaudric M, Rohof WO, Smout AJ, Tack J, Zwinderman AH, Zaninotto G, Busch OR; European Achalasia Trial Investigators. Pneumatic dilation versus laparoscopic Heller's myotomy for idiopathic achalasia. N Engl J Med. 2011 May 12;364(19):1807-16. doi: 10.1056/NEJMoa1010502. PMID 21561346
- See also: Homepage of Nanfang Hospital of Southern Medical University — http://www.nfyy.com/
- See also: Homepage of Department of Gastroenterology, Nanfang Hospital of Southern Medical University — http://www.xhbnet.com/